CLINICAL TRIAL: NCT03741231
Title: 18FluoroDeoxyGlucose-Positron Emission Tomography (PET) in Patients With Melanoma or Non Small Cell Lung Cancer Treated With Immunotherapy
Brief Title: 18FDG-PET in Patients With Melanoma or NSCLC Treated With Immunotherapy
Acronym: IMMUNOPET
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: IMMUNOPET ( 29BRC17.0253).
Record Dates: First submitted 2018-07-13; First posted 2018-11-14 (Actual); Last update posted 2019-05-06 (Actual); Status verified 2019-03

CONDITIONS: Melanoma; NSCLC; Positron-Emission Tomography; Immunotherapy; 18F-FDG
Keywords: melanoma; NSCLC; FDG; PET; immunotherapy
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Study the EFS and OS according to 18FDG PET in patients with melanoma or non small cell lung cancer treated by immunotherapy.

DETAILED DESCRIPTION:
Study EFS in patients with melanoma or NSCLC treated by immunotherapy (anti CTLA4 or anti PDL1) and performed18FDG PET

Multicentric retrospective study

ELIGIBILITY:
Inclusion Criteria:

* patients treated for melanoma or NSCLC with immunotherapy (anti CTLA4 or antiPDL1)
* patients treated in Brest, Morlaix, Landerneau hospital
* patients performed FDG PET
* no opposition to study

Exclusion Criteria:

* age under 18 years old
* refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 70 patients (50 patients with melanoma and 20 patients with NSCLC)
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
measure of progression free survival (obtained by the delay between the date of initiation of immunotherapy until the date of first documented progression disease in patients with melanoma or NSCLC treated by immunotherapy | up to 50 months
  From date of initiation of treatment until the date of first documented progression disease according to different criteria in interim PET/CT 1.
  18F-FDG PET/CT imaging was performed prior to (18F-FDG PET/CT 0) and 14 weeks after ICI onset (18F-FDG PET/CT 1). Assessment of patient response to treatment was done according to RECIST1.1, iRECIST, PERCIST and PECRIT criteria.

SECONDARY OUTCOMES:
measure of overall survival (obtained by the delay between the date of initiation of immunotherapy until the date of death related to disease in patients with melanoma or NSCLC treated by immunotherapy | up to 50 months
  From date of initiation of treatment until the date of death related to disease according to different criteria in interim PET/CT 1.
  18F-FDG PET/CT imaging was performed prior to (18F-FDG PET/CT 0) and 14 weeks after ICI onset (18F-FDG PET/CT 1). Assessment of patient response to treatment was done according to RECIST1.1, iRECIST, PERCIST and PECRIT criteria.
Study different criteria (RECIST, iRECIST, PERCIST and PECRIT) to predict PFS or OS | up to 50 months
  Interpretation according to 4 criteria to predict response to immunotherapy
study the potential correlation between PET data and clinicobiological data | up to 50 months
  correlation between adverse events (AE) due to immunotherapy described on PET data and AE detected on clinicobiological data

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - CHRU de Brest, Brest
  - CH de LANDERNEAU, Landerneau
  - Centre Hospitalier de Morlaix, Morlaix